CLINICAL TRIAL: NCT07351890
Title: Study on the Diagnostic Accuracy of Endoscopic Ultrasound for Submucosal Masses of Colorectal Cancer
Brief Title: Diagnostic Accuracy of EUS for Colorectal Submucosal Masses
Status: Completed | Type: Observational
Sponsor: Run-hua Li (Other)
Responsible Party: Sponsor-Investigator, Run-hua Li, Study Director, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Other Study IDs: NYSZYYEC20230088
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Subepithelial Lesions
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endoscopic Ultrasound (EUS) Assessment

SUMMARY:
This study aims to evaluate the diagnostic accuracy of endoscopic ultrasound (EUS) for colorectal submucosal tumors/lesions (SMTs/SELs) and to identify factors associated with correct EUS diagnosis. Using cases with histopathologic confirmation as the reference standard, EUS-based preoperative diagnoses will be compared with final pathology to estimate overall accuracy and accuracy across different lesion types. Potential influencing factors-including lesion location, size, echogenicity, layer of origin, image quality, operator experience and training, and EUS equipment/probe type-will be analyzed to determine independent predictors of diagnostic concordance. The findings are expected to inform optimization of EUS examination and interpretation for colorectal submucosal lesions, thereby improving clinical decision-making and overall quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted to Shenzhen Hospital of Southern Medical University from 2015 to 2023 and underwent colorectal endoscopic ultrasound.
* Patients diagnosed with colorectal submucosal tumors (subepithelial lesions) according to the Chinese expert consensus on the endoscopic diagnosis and treatment of gastrointestinal submucosal tumors (2023 edition).

Exclusion Criteria:

* Patients with endoscopic ultrasound diagnosis of non-submucosal tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients who were admitted to Shenzhen Hospital of Southern Medical University between 2015 and 2023 and underwent colorectal endoscopic ultrasound (EUS). Eligible participants are those diagnosed with colorectal submucosal tumors/subepithelial lesions based on the Chinese expert consensus on endoscopic diagnosis and treatment of gastrointestinal submucosal tumors (2023 edition) and related criteria. Patients whose EUS findings did not support a diagnosis of a submucosal tumor/subepithelial lesion were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Coincidence Rate Between Endoscopic Ultrasound Diagnosis and Pathological Diagnosis | At the time of preoperative EUS and postoperative pathological evaluation (Day 0).
  For each included lesion with histopathologic confirmation, the preoperative endoscopic ultrasound (EUS) diagnosis will be compared with the final pathological diagnosis. The coincidence rate will be calculated as the proportion of lesions in which the EUS diagnosis is concordant with the pathological diagnosis (number of concordant diagnoses divided by the total number of lesions assessed) during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://rs.yiigle.com/cmaid/1460987

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT07351890/Prot_SAP_000.pdf